CLINICAL TRIAL: NCT00872677
Title: A Culturally-Tailored Weight Loss Program
Brief Title: Weight Loss Counseling for African American Women Who Are Breast Cancer Survivors
Status: Completed | Type: Observational
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000612147; 013003B3E (Other: Wayne State University - Human Investigation Committee); NCT00082056 (obsolete NCT alias)
Record Dates: First submitted 2009-03-28; First posted 2009-03-31 (Estimated); Last update posted 2013-04-29 (Estimated); Status verified 2013-04

CONDITIONS: Breast Cancer; Obesity; Weight Changes
Keywords: weight changes; obesity; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms; Obesity; Body Weight Changes | interventions — Diet

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Dietitian-led counseling and Weight Watchers: Talk to study dietitian (eight in person or by phone) weekly for the first 3 months, every other week for the next 3 months and monthly thereafter.
  Interventions: Behavioral: Diet
- Dietitian & Weight Watchers + Spirituality Counseling: Dietitian wkly for the 1st-3 months, every other week for the next 3 months and monthly thereafter; Spiritual counselor weekly in months 6-9, every other week in months 9-12 and monthly thereafter.
  Interventions: Behavioral: Diet; Other: Spiritual counseling

INTERVENTIONS:
Behavioral: Diet — Talk to study dietitian (eight in person or by phone) weekly for the first 3 months, every other week for the next 3 months and monthly thereafter.
Other: Spiritual counseling — Spiritual counselor weekly in months 6-9, every other week in months 9-12 and monthly thereafter.
  Groups: Dietitian & Weight Watchers + Spirituality Counseling

SUMMARY:
RATIONALE: A culturally sensitive weight loss program for obese African American breast cancer survivors may be more effective than a standard weight loss program in helping women lose weight.

PURPOSE: This randomized clinical trial is studying personalized weight loss counseling to see how well it works in African American women who are breast cancer survivors.

DETAILED DESCRIPTION:
OBJECTIVES:

* To develop a weight loss intervention for obese African American women who are breast cancer survivors.

OUTLINE: This is a randomized study. Participants are randomized to 1 of 2 intervention groups.

* Group 1: Participants receive traditional individual dietary and exercise counseling in combination with the Weight Watchers weight loss program for 18 months.
* Group 2: Participants receive individual dietary and exercise counseling in combination with the Weight Watchers weight loss program as in group 1. They also receive spiritual counseling that incorporates meditation, readings, and the recording of thoughts into a long-term weight management program. The program addresses coping with stress, setting priorities, dealing with emotional issues that trigger old behavior patterns, and developing accountability for following desired diet and exercise patterns.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of breast cancer within the past 5 years

  * Stage I-IIIA disease
  * No recurrence of cancer
* Identified as African American
* Body Mass Index 30-40
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* Stable body weight
* Not currently following a special diet
* No uncontrolled congestive heart failure, untreated hypertension, disabling osteoarthritis, drug or alcohol abuse, or psychiatric conditions that may interfere with counseling

PRIOR CONCURRENT THERAPY:

* More than 3 months since prior chemotherapy or radiotherapy

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Two groups to participate:
  Group 1: Dietitian led counseling and Weight Watchers groups for 18 months Group 2: Dietitian led counseling and Weight Watchers groups for 18 months with Spirituality counseling from 6 to 18 months.
Sampling Method: Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2004-05; Primary Completion 2006-10 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Weight change | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael S. Simon, MD, MPH, Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States

REFERENCES:
- [Result] Djuric Z, Mirasolo J, Kimbrough L, Brown DR, Heilbrun LK, Canar L, Venkatranamamoorthy R, Simon MS. A pilot trial of spirituality counseling for weight loss maintenance in African American breast cancer survivors. J Natl Med Assoc. 2009 Jun;101(6):552-64. doi: 10.1016/s0027-9684(15)30940-8. PMID 19585923